CLINICAL TRIAL: NCT06466798
Title: Fourth Ventricular Administration of Immune Checkpoint Inhibitor (Nivolumab) and Methotrexate or 5-Azacytidine for Recurrent Medulloblastoma, Ependymoma, and Other CNS Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to find participants meeting eligibility critieria
Sponsor: Jeffrey Treiber (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Treiber, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-0240
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Ependymoma; Recurrent Medulloblastoma; CNS Malignancies
MeSH Terms: conditions — Ependymoma; Medulloblastoma; Central Nervous System Neoplasms | interventions — Nivolumab; Methotrexate; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab plus Methotrexate (Experimental): Enrolled patients with medulloblastoma and other CNS malignancies will receive:
  1. Intraventricular Methotrexate infusions 2 mg daily for 4 consecutive days per week every other week on weeks 1, 3, 5, 7, 9, and 11.
  2. Intraventricular Nivolumab infusions. Nivolumab will be administered once every other week on weeks 2, 4, 6, 8, 10, and 12. Dosing will be based upon patient body weight.
  Interventions: Drug: Nivolumab; Drug: Methotrexate
- Nivolumab plus 5-Azacytidine (Experimental): Enrolled patients with ependymoma will receive:
  1. Intraventricular 5-Azacytidine infusions 10 mg once weekly for twelve consecutive weeks.
  2. Intraventricular Nivolumab infusions once every other week on weeks 1, 3, 5, 7, 9, and 11. Dosing will be based upon patient body weight.
  Interventions: Drug: Nivolumab; Drug: 5-Azacytidine

INTERVENTIONS:
Drug: Nivolumab — Nivolumab infusions will be given intraventricularly once every other week for 12 weeks. Dosing will be based upon patient body weight.
Drug: Methotrexate — 2 mg methotrexate infusions will be given intraventricularly daily for 4 consecutive days per week every other week for 12 weeks.
  Arms: Nivolumab plus Methotrexate
Drug: 5-Azacytidine — 10 mg 5-Azacytidine infusions will be given intraventricularly once weekly for twelve consecutive weeks.
  Arms: Nivolumab plus 5-Azacytidine

SUMMARY:
The goal of this clinical trial is to assess the safety, toxicity, and antitumor activity of fourth ventricular infusions of nivolumab plus 5-azacytidine for recurrent ependymoma and nivolumab plus methotrexate for recurrent medulloblastoma and other CNS malignancies.

Additionally, the study will explore immunologic responses to nivolumab.

The hypothesis is that local administration of nivolumab, an immune checkpoint inhibitor, is safe and will lead to even more robust treatment responses when administered following 5-azacytidine in patients with recurrent ependymoma or methotrexate in patients with medulloblastoma or other CNS tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 - 80 years at time of recurrence or progression
* Minimum body weight of 10 kilograms
* Diagnosis: Patients with histologically verified medulloblastoma, ependymoma, with recurrence or progression anywhere in the brain and/or spine. Patients are also eligible if they have refractory disease, which will be defined as residual tumor which has not been completely cleared despite prior treatments. To be eligible, patients' disease must have originated or recurred in the posterior fossa of the brain. Patients with central nervous system (CNS) malignancies besides medulloblastoma and ependymoma are also eligible if they have recurrent or refractory disease in the posterior fossa
* Patient must have either measurable or evaluable tumor as assessed by magnetic resonance imaging (MRI) of the brain and total spine. If the patient does not have measurable or evaluable tumor after surgery for resection and catheter placement, infusions will be held until there is measurable or evaluable tumor on subsequent MRI scans. Patients with no measurable or evaluable disease after surgical resection cannot receive other systemic or intraventricular therapies and remain on study. If patients or their guardians choose to pursue additional systemic or intraventricular therapies during this time, the patients will be removed from the study. If patients do not receive additional systemic or intraventricular therapies and the is measurable or evaluable disease on subsequent imaging studies, then infusions may proceed according to the study protocol.
* An implanted catheter in the fourth ventricle or posterior fossa tumor cavity attached to a ventricular access device or agreement to have one placed.
* Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea
* For patients receiving biologic or investigational agents (anti-neoplastic), the last dose must have been received at least 7 days prior to study enrollment. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which such events are known to occur
* For patients receiving monoclonal antibody treatment and agents with prolonged half-lives, the last dose of the agent must have been received at least 28 days prior to study enrollment
* For patients receiving Immune Effector Cell (IEC) Therapy (e.g., Chimeric antigen receptor (CAR) T-cells), viral therapy, or cellular therapy, patients must have received therapy ≥ 3 months prior to study enrollment. Patients who have received allogeneic stem cell transplants must wait at least 6 months prior to enrollment with no evidence of active graft versus host disease. Patients who have received autologous stem cell transplants must wait at least 3 months since transplant to enroll.
* Patients must have received their last fraction of standard upfront radiation ≥ 3 months prior to enrollment and ≥ 28 days for palliative radiation.
* Life expectancy of at least 12 weeks in the opinion of the principal investigator
* Lansky score of 50 or greater if ≤16 years of age or Karnofsky score of 50 or greater if > 16 years of age
* Patients must have recovered from the acute toxic effects of all prior anticancer chemotherapy
* Patients must have adequate organ and marrow function as defined below:
* Absolute neutrophil count > 1.0 x 10^9 cells/L
* Platelets > 50 x 10^9 cells/L (unsupported, defined as no platelet transfusion within 7 days)
* Hemoglobin ≥ 8 g/dL (may receive transfusions)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* prothrombin time test with an international normalized ratio (PT/INR), partial thromboplastin time (PTT) ≤ 1.5 x ULN
* Alanine aminotransferase (ALT) [serum glutamic-pyruvic transaminase (SGPT)] and aspartate aminotransferase (AST) [serum glutamic-oxaloacetic transaminase (SGOT)] < 3 x institutional upper limit of normal (ULN)
* Albumin ≥ 3 g/dL
* Normal creatinine level for age according to hospital or outside lab standards. If creatinine is outside normal range, then Chronic kidney disease (CKD)-epi calculation will be performed for patients age >25. Patients age > 25 with estimated glomerular filtration rate (eGFR) > 60 ml/min/1.73m2 will be eligible and patients who do not meet this standard require nephrologist consultation to determine safety of enrollment. For patients ages 1 to 25 with creatinine outside normal range, Chronic kidney disease (CKD)--U25 calculation will be performed. Patients ages 1 to 25 with eGFR > 40 ml/min/1.73m2 will be eligible and patients who do not meet this standard require nephrologist consultation to determine safety of enrollment.
* Patient or patient's legal representative, parent(s), or guardian able to provide written informed consent.
* Patients of childbearing age and their parents will be informed that pregnancy is an exclusion criterion for the study. Male patients will be informed to use condoms if sexually active. Female patients will be advised to use contraceptives to prevent pregnancy if sexually active including male or female condoms, oral contraceptives, contraceptive injections, or other forms of contraception advised by primary care physician or obstetrician/gynecologist

Exclusion Criteria:

* Enrolled in another treatment protocol
* Patient is currently receiving corticosteroids that cannot be weaned off at least one week prior to first Nivolumab infusion
* Evidence of untreated infection
* Pregnant or lactating women
* Patient that has had allogenic stem cell transplant

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the number of participants with a new neurological toxicity that is graded as Grade 3 or higher and that is probably or definitely related to infusions [that is, classified as dose-limiting toxicity (DLT)] | from start of treatment to end of treatment (about 12 weeks)
  Adverse events will be graded according to the NCI common terminology criteria version 5.0. Adverse events not included in the Common Terminology Criteria for Adverse Events (CTCAE) chart will be graded as follows:
  * Grade 1: Mild: discomfort present with no disruption of daily activity, no treatment required beyond prophylaxis
  * Grade 2: Moderate: discomfort present with some disruption of daily activity, require treatment.
  * Grade 3: Severe: discomfort that interrupts normal daily activity, not responding to first line treatment.
  * Grade 4: Life Threatening: discomfort that represents immediate risk of death.

SECONDARY OUTCOMES:
Number of participants who responded to therapy as determined by MRI imaging | baseline, within 7 days of completing final infusion (about 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Treiber, MD, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: No